CLINICAL TRIAL: NCT00256867
Title: A 16 Week Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of a New Medication (GSK523338) to Lower LDL-c and HbA1c in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study In Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: AVS101946
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK523338

SUMMARY:
This study evaluates the effect of medicines for type 2 diabetes and lipids control. This study will require about 6 office visits for lab tests and examinations. All study related medicines and medical examinations will be provided at no cost to the subjects.

ELIGIBILITY:
Inclusion criteria:

* A clinical diagnosis type 2 diabetes mellitus.
* Women must not be pregnant or breastfeeding during the study and 30 days after the study.
* Must sign an informed consent form at the study clinic.

Exclusion criteria:

* Severe chronic diseases that would prevent from participating and completing the study by investigator's judgement.
* Use of an investigational drug within 30 days or 5 half lives before first dose of study medication.
* Insulin use for > 1 week in past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2005-08-18 (Actual); Primary Completion 2006-10-31 (Actual); Study Completion 2006-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (78):
- United States (41):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Waltham, Massachusetts
  - GSK Investigational Site, City of Saint Peters, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Jamaica, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Tualatin, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Clinton, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Vancouver, Washington
- Australia (8):
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Keswick, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Heidelberg West, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
- Canada (22):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Mount Pearl, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Granby, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Plessisville, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- GSK Investigational Site, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVS101946 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 17 April 2005 and 21 December 2006 at 68 centers in five countries including United States, Canada, Australia, Mexico, and the Philippines. A total of 370 participants were randomized of which 1 participant did not received study medication remaining 369 participants were included in safety population.
Pre-assignment Details: Out of the 369 participants from safety population, 12 participants received at least one dose but did not have at least one On-Therapy value for any efficacy assessment, the remaining 357 participants were included in Intent- to-Treat population.
Groups:
- Fixed Dose Combination (FDC) 4/40 Milligram (mg): Participants received FDC of rosiglitazone (RSG) 4.0 mg and simvastatin (SIMV) 40 mg (FDC 4/40) and matching placebo once a day for 16 weeks. In case of the participants who had Low Density Lipoprotein-cholesterol (LDL-c) > 130 milligram per deciliter (mg/dL) at Visit 4a (Week 6) the treatment doses were up titrated to FDC RSG/SIMV 4/40 mg and SIMV 40 mg from Week 6 till Week 16.
- FDC 4/80 mg: Participants received FDC RSG/SIMV 4/80 mg and SIMV 40 mg matching placebo once a day for 16 weeks.
- FDC 8/40 mg: Participants received FDC RSG/SIMV 8/40 mg once a day and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to FDC RSG/SIMV 8/40 mg and SIMV 40 mg from Week 6 till Week 16.
- FDC 8/80 mg: Participants received FDC RSG/SIMV 8/80 mg and matching placebo once a day for 16 weeks.
- RSG 4mg: Participants received RSG 4.0 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL evaluated at Visit 4a (Week 6), the treatment doses were titrated up to RSG/SIMV 4/40 mg once a day from Week 6 till Week 16.
- RSG 8mg: Participants received RSG 8.0 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to RSG/SIMV 8/40 mg once a day from Week 6 till Week 16.
- SIMV 40mg: Participants received SIMV 40 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to SIMV/SIMV 40/40 mg once a day from Week 6 till Week 16.
- SIMV 80mg: Participants received SIMV/SIMV 40/40 mg once a day for 16 weeks.
Period: Overall Study
Arm/Group | Fixed Dose Combination (FDC) 4/40 Milligram (mg) | FDC 4/80 mg | FDC 8/40 mg | FDC 8/80 mg | RSG 4mg | RSG 8mg | SIMV 40mg | SIMV 80mg
Started | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47
Completed | 45 | 39 | 40 | 40 | 41 | 40 | 41 | 36
Not Completed | 2 | 5 | 5 | 6 | 7 | 6 | 5 | 11
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 2 | 2 | 3 | 2 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 2
Not completed — Fasting plasma glucose >240 mg/dL | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Glycemia over 13.3 millimole per litre | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator's Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance with study medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant travelled Overseas | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant out of assessment window | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by participant | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all participants who were randomized and received at least one dose of study medication. No race information available for one participant in arm SIMV 40mg.
Groups:
- FDC RSG/SIMV 4/40 mg: Participants received FDC RSG/SIMV 4/40 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6), the treatment doses were up titrated to FDC RSG/SIMV 4/40 mg and SIMV 40 mg once a day from Week 6 till Week 16.
- FDC RSG/SIMV 4/80 mg: Participants received FDC RSG/SIMV 4/80 mg and SIMV 40 mg matching placebo once a day for 16 weeks.
- FDC RSG/SIMV 8/40 mg: Participants received FDC RSG/SIMV 8/40 mg once a day and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to FDC RSG/SIMV 8/40 mg and SIMV 40 mg once a day from Week 6 till Week 16.
- FDC RSG/SIMV 8/80 mg: Participants received FDC RSG/SIMV 8/80 mg and matching placebo once a day for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4mg | RSG 8mg | SIMV 40mg | SIMV 80mg | Total
Number analyzed (Participants) | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47 | 369
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (9.13) | 55.1 (10.31) | 56.9 (9.07) | 55 (8.65) | 53.8 (11.37) | 54.6 (9.93) | 53.4 (9.03) | 53.5 (10.49) | 54.6 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 23 | 22 | 24 | 25 | 25 | 25 | 190
  Male | 24 | 21 | 22 | 24 | 24 | 21 | 21 | 22 | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 0 | 5 | 6 | 7 | 3 | 2 | 2 | 26
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian - Central/South Asian Heritage | 1 | 4 | 4 | 1 | 4 | 2 | 3 | 4 | 23
  Asian - East Asian Heritage | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 5
  Asian - South East Asian Heritage | 10 | 6 | 12 | 6 | 7 | 5 | 10 | 11 | 67
  Native Hawaiian or other Pacific Islander | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White - Arabic/North African Heritage | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 2 | 8
  White -White/Caucasian/European Heritage | 28 | 23 | 20 | 30 | 27 | 27 | 28 | 20 | 203
  Mixed Race | 4 | 7 | 1 | 1 | 2 | 8 | 2 | 6 | 31
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change From Baseline to Week 6 in LDL-c in FDC and RSG Monotherapy
Description: Median percent change from Baseline to Week 6 in LDL-c in FDC and RSG monotherapy was reported. Percent change from Baseline = 100*(exponent [change on log scale]-1). Baseline assessments were recorded at Visit 3 (Week 0). For a missing Baseline value, the Baseline value were replaced by the last pre-treatment measurement, if available. The hypothesis of treatment difference was tested at a 0.05 significance level based on two-sided tests. The point estimates and corresponding 95% confidence intervals for treatment differences was calculated. Treatment differences were assessed within the context of an analysis of covariance (ANCOVA) with terms for treatment, gender, current sulfonylurea use (at baseline), country, and Baseline measurement. ANCOVA for LDL-c were performed based on log-transformed data.
Time Frame: Baseline (Week 0) and Week 6
Population: Intent-to-Treat Population comprised of all participants who were randomized and had at least one On-Therapy value for an efficacy assessment. The Intent-to-Treat population with last observation carried forward (LOCF) was used for efficacy analyses. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Percent change in LDL-c
Groups:
- All FDC RSG/SIMV Groups: In this arm, all the participants were pooled who received FDC RSG/SIMV 4/40 mg, FDC RSG/SIMV 4/80 mg, FDC RSG/SIMV 8/40 mg, FDC RSG/SIMV 8/80 mg and matching placebo once a day for 16 weeks.
- All RSG Monotherapy Groups: In this arm, all the participants were pooled who received RSG 4 and 8mg, and matching placebo once a day for 16 weeks.
Arm/Group | All FDC RSG/SIMV Groups | All RSG Monotherapy Groups
Number analyzed (Participants) | 171 | 88
Percent change in LDL-c | -39.9 [-69 to 56] | 5.4 [-31 to 67]
Statistical Analysis 1: Comparison: All FDC RSG/SIMV Groups vs All RSG Monotherapy Groups; Test type: Superiority or Other; p < 0.0001, ANCOVA; Ratio Expressed as percent difference = -37.186, 95% CI 2-sided [-41.219 to -32.879] — Estimation parameter was Ratio to RSG Group expressed as percent difference from RSG group. Based on ANCOVA : Log(value) - log(baseline)= log(baseline) + sex + country + Treatment + Prior Sulfonylurea use

2. Secondary Outcome: Mean Change From Baseline to Week 16 in Glycosylated Hemoglobin A1c (HbA1c) in FDC and SIMV Monotherapy
Description: Mean change from Baseline to Week 16 in HbA1c in FDC and SIMV monotherapy was reported. Change from Baseline was computed as (Visit value - Baseline value). Baseline assessments were recorded at Visit 3 (Week 0). For a missing Baseline value, the Baseline value were replaced by the last pre-treatment measurement, if available. The hypothesis of treatment difference was tested at a 0.05 significance level based on two-sided tests. The point estimates and corresponding 95% confidence intervals for treatment differences was calculated. Treatment differences were assessed within the context of ANCOVA with terms for treatment, gender, current sulfonylurea use (at Baseline), country, and Baseline measurement.
Time Frame: Baseline (Week 0) and Week 16
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- All SIM Monotherapy Groups: In this arm, all the participants were pooled who received SIM 40 and 80 mg, and matching placebo once a day for 16 weeks.
Arm/Group | All SIM Monotherapy Groups | All FDC RSG/SIMV Groups
Number analyzed (Participants) | 90 | 176
mg/dL | -0.01 (1.131) | -0.83 (1.093)
Statistical Analysis 1: Comparison: All SIM Monotherapy Groups vs All FDC RSG/SIMV Groups; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.09 to -0.55] — Change = Baseline + sex + country + Treatment + Prior Sulfonylurea use

3. Secondary Outcome: Median Percent Change From Baseline to Week 6 in LDL-c
Description: Percent change from Baseline = 100*(exponent [change on log scale]-1). Baseline assessments were recorded at Visit 3 (Week 0). For a missing Baseline value, the Baseline value were replaced by the last pre-treatment measurement, if available.
Time Frame: Baseline (Week 0) and Week 6
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Percent change in LDL-c
Groups:
- RSG 4 mg: Participants received RSG 4.0 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL evaluated at Visit 4a (Week 6), the treatment doses were titrated up to RSG/SIMV 4/40 mg once a day from Week 6 till Week 16.
- RSG 8 mg: Participants received RSG 8.0 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to RSG/SIMV 8/40 mg once a day from Week 6 till Week 16.
- SIMV 40 mg: Participants received SIMV 40 mg and matching placebo once a day for 16 weeks. In case of the participants who had LDL-c >130 mg/dL at Visit 4a (Week 6) the treatment doses were up titrated to SIMV/SIMV 40/40 mg once a day from Week 6 till Week 16.
- SIMV 80 mg: Participants received SIMV/SIMV 40/40 mg once a day for 16 weeks.
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 44 | 42 | 40 | 45 | 47 | 41 | 42 | 46
Percent change in LDL-c | -32.7 [-62 to 39] | -39.4 [-67 to 56] | -39.0 [-64 to 17] | -44.4 [-69 to 18] | 5.6 [-31 to 67] | 5.4 [-26 to 62] | -34.0 [-65 to 75] | -44.2 [-73 to 28]

4. Secondary Outcome: Mean Change From Baseline to Week 16 in HbA1c
Description: Change from Baseline was computed as (Visit value - Baseline value). Baseline assessments were recorded at Visit 3 (Week 0). For a missing Baseline value, the Baseline value were replaced by the last pre-treatment measurement, if available.
Time Frame: Baseline (Week 0) and Week 16
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 45 | 44 | 42 | 45 | 46 | 43 | 43 | 47
mg/dl | -0.52 (0.966) | -0.54 (1.285) | -1.24 (1.035) | -1.06 (0.901) | -1.04 (0.964) | -1.31 (1.216) | 0.00 (0.989) | -0.02 (1.258)

5. Secondary Outcome: Mean Change From Baseline to Week 16 in Fasting Plasma Glucose (FPG)
Description: as for outcome 4
Time Frame: Baseline (Week 0) and Week 16
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimol per litre (mmol/L)
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 45 | 43 | 42 | 45 | 47 | 43 | 43 | 46
Millimol per litre (mmol/L) | -0.31 (2.202) | -1.29 (3.365) | -2.10 (2.018) | -1.90 (2.176) | -1.88 (2.386) | -2.23 (1.621) | 0.43 (2.526) | 0.37 (2.483)

6. Secondary Outcome: Number of Participant With LDL<100 mg/dL (2.59 mmol/L) at Week 6
Description: Number of participants achieving American Diabetes Association (ADA) target of LDL<100 mg/dL (2.59 mmol/L) at Week 6 was compared between the FDC groups and the all SIMV group using logistic regression with terms for treatment, Baseline value, gender and current sulfonylurea use (at Baseline) in the model.
Time Frame: Week 6
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All RSG Monotherapy Groups | All FDC RSG/SIMV Groups
Number analyzed (Participants) | 88 | 171
Participants | 20 | 148
Statistical Analysis 1: Comparison: All RSG Monotherapy Groups vs All FDC RSG/SIMV Groups; Test type: Superiority or Other; p < .0001, ANCOVA; Odds Ratio (OR) = 36.32, 95% CI [16.52 to 79.85] — Odds (logistic regression:log odds=Baseline + sex + Treatment + Prior Sulfonylurea use) of having an LDL-c < 100 mg/dL at Week 6 on All FDC RSG/SIMV groups compared to All RSG monotherapy groups

7. Secondary Outcome: Number of Participants With HbA1c < 7.0% or Reduction of HbA1c ≥ 0.7% at Week 16
Description: Number of participants achieving ADA target of HbA1c < 7.0% or reduction of HbA1c ≥ 0.7% at Week 16 was compared between the FDC groups and the RSG groups groups using logistic regression with terms for treatment, Baseline value, gender and current sulfonylurea use (at Baseline) in the model.
Time Frame: Up to Week 16
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All SIM Monotherapy Groups | All FDC RSG/SIMV Groups
Number analyzed (Participants) | 90 | 176
Participants | 26 | 108
Statistical Analysis 1: Comparison: All SIM Monotherapy Groups vs All FDC RSG/SIMV Groups; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 4.05, 95% CI 2-sided [2.32 to 7.07] — Odds (logistic regression: log odds=Baseline + sex + Treatment + Prior SU use) of having an HbA1c < 7% or reduction of HbA1c >= 0.7% at Week 16 on All FDC group compared to Simv group

8. Secondary Outcome: Number of Participants With FPG< 126 mg/dL (7.0 mmol/L) or Reduction of FPG ≥ 30 mg/dL (1.67 mmol/L) at Week 16
Description: Number of participants achieving ADA target of FPG< 126 mg/dL (7.0 mmol/L) or reduction of FPG ≥ 30 mg/dL (1.67 mmol/L) at Week 16 was compared between the all SIM monotherapy group and the all FDC RSG/SIMV groups using logistic regression with terms for treatment, Baseline value, gender and current sulfonylurea use (at Baseline) in the model.
Time Frame: Week 16
Population: Intent-to-Treat with LOCF. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All SIM Monotherapy Groups | All FDC RSG/SIMV Groups
Number analyzed (Participants) | 89 | 175
Participants | 22 | 96
Statistical Analysis 1: Comparison: All SIM Monotherapy Groups vs All FDC RSG/SIMV Groups; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 3.93, 95% CI 2-sided [2.21 to 7] — Odds (logistic regression:log odds=Baseline + sex + Treatment + Prior SU use) of having an FPG < 7.0 mmol/L or reduction of FPG >= 1.67 mmol/L at Week 16 on All FDC group compared to Simv group

9. Secondary Outcome: On-Therapy Vital Signs of Potential Clinical Concern Including Systolic, Diastolic Blood Pressure and Heart Rate
Description: The potential clinical importance ranges (low and high) of the vital sign parameters were for systolic blood pressure (<85 and >160 millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to Week 16
Population: Safety Population comprised of all participants who were randomized and received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 45 | 44 | 42 | 45 | 47 | 43 | 43 | 46
Participants
  Systolic BP, High | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0
  Systolic BP, Low | 0 | 0 | 2 | 3 | 2 | 3 | 0 | 1
  Diastolic BP, High | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Diastolic BP, Low | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Heart Rate, Low | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2

10. Secondary Outcome: On-Therapy Change From Baseline in Body Weight
Description: Baseline assessments were recorded at Visit 3 (Week 0). For a missing Baseline value, the Baseline value were replaced by the last pre-treatment measurement, if available. Change from Baseline was computed as: Visit value - Baseline Value.
Time Frame: Up to Week 16
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47
Kilogram
  Week 6: number analyzed (Participants) | 45 | 44 | 42 | 45 | 47 | 42 | 43 | 46
  Week 6 | 0.9 (3.45) | -0.3 (2.83) | 0.0 (1.80) | 0.4 (1.85) | 0.5 (2.07) | 0.8 (2.66) | -0.5 (1.84) | -0.2 (1.93)
  Week 16: number analyzed (Participants) | 45 | 41 | 39 | 42 | 40 | 40 | 42 | 37
  Week 16 | 0.4 (4.39) | 0.8 (2.75) | 1.7 (2.51) | 1.1 (3.98) | 1.4 (4.41) | 2.2 (3.94) | -0.5 (3.26) | -1.5 (3.57)

11. Secondary Outcome: Number of Participants With Specified Ranges of Red and White Blood Cell Counts Detected in Urine
Description: Urine samples were observed for red blood cells and white blood cells. the results were reported as cells per high-power field (cells/HPF). The number of participants with cells in urine were reported.
Time Frame: Up to Week 16
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47
Participants
  0-1, Red Blood Cells/HPF | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 2
  1-3, Red Blood Cells/HPF | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 1
  10-15, Red Blood Cells/HPF | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  15-25, Red Blood Cells/HPF | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  3-5, Red Blood Cells/HPF | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  5-10, Red Blood Cells/HPF | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
  50-100, Red Blood Cells/HPF | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  None seen, Red Blood Cells/HPF | 6 | 3 | 8 | 8 | 9 | 8 | 7 | 12
  0-1, White Blood Cells/HPF | 2 | 1 | 3 | 5 | 3 | 4 | 2 | 4
  1-3, White Blood Cells/HPF | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  10-15, White Blood Cells/HPF | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  15-25, White Blood Cells/HPF | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
  25-50, White Blood Cells/HPF | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  3-5, White Blood Cells/HPF | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  5-10, White Blood Cells/HPF | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 3
  50-100, White Blood Cells/HPF | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Innumerable, White Blood Cells/HPF | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  None seen, White Blood Cells/HPF | 3 | 2 | 6 | 3 | 6 | 5 | 7 | 6

12. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Event (SAE)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to Week 16
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47
Participants
  Any AEs | 21 | 23 | 22 | 26 | 19 | 25 | 23 | 21
  Any SAEs | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0

13. Secondary Outcome: Number of of Participants With Laboratory Evaluations of Potential Clinical Concern at Any Time Post-baseline
Description: The clinical chemistry parameters analyzed were sodium, potassium, bicarbonate, chloride, calcium, total protein, albumin, creatinine total bilirubin, blood urea nitrogen, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transpeptidase, and alkaline phosphatase. The hematology parameters analyzed were hemoglobin, hematocrit, platelet count, total white cell count. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important hematology findings at any visit were reported.
Time Frame: Up to Week 16
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
Number analyzed (Participants) | 47 | 44 | 45 | 46 | 48 | 46 | 46 | 47
Participants
  Hematocrit, Low: number analyzed (Participants) | 45 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Hematocrit, Low | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 0
  Hemoglobin, Low: number analyzed (Participants) | 45 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Hemoglobin, Low | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 3
  White Blood Cells count, Low: number analyzed (Participants) | 45 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  White Blood Cells count, Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Platelet Count, High: number analyzed (Participants) | 45 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Platelet Count, High | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Alanine Amino Transferase, High: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Alanine Amino Transferase, High | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate Amino Transferase, High: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Aspartate Amino Transferase, High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Carbon Dioxide content / Bicarbonate, Low: number analyzed (Participants) | 46 | 44 | 44 | 45 | 46 | 46 | 44 | 46
  Carbon Dioxide content / Bicarbonate, Low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatine Kinase, High: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Creatine Kinase, High | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gamma Glutamyl Transferase, High: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Gamma Glutamyl Transferase, High | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1
  Calcium, Low: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Calcium, Low | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium, High: number analyzed (Participants) | 46 | 44 | 44 | 45 | 48 | 46 | 44 | 46
  Potassium, High | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and nSAEs were recorded up to Week 16
Description: Safety population was used to record AEs
Arm/Group | FDC RSG/SIMV 4/40 mg | FDC RSG/SIMV 4/80 mg | FDC RSG/SIMV 8/40 mg | FDC RSG/SIMV 8/80 mg | RSG 4 mg | RSG 8 mg | SIMV 40 mg | SIMV 80 mg
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44 | 0/42 | 0/45 | 0/47 | 0/43 | 0/44 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/44 | 1/45 | 1/46 | 0/48 | 3/46 | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 4/47 | 4/44 | 3/45 | 10/46 | 4/48 | 4/46 | 5/46 | 6/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDC RSG/SIMV 4/40 mg (N=47) | FDC RSG/SIMV 4/80 mg (N=44) | FDC RSG/SIMV 8/40 mg (N=45) | FDC RSG/SIMV 8/80 mg (N=46) | RSG 4 mg (N=48) | RSG 8 mg (N=46) | SIMV 40 mg (N=46) | SIMV 80 mg (N=47)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC RSG/SIMV 4/40 mg (N=47) | FDC RSG/SIMV 4/80 mg (N=44) | FDC RSG/SIMV 8/40 mg (N=45) | FDC RSG/SIMV 8/80 mg (N=46) | RSG 4 mg (N=48) | RSG 8 mg (N=46) | SIMV 40 mg (N=46) | SIMV 80 mg (N=47)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.